CLINICAL TRIAL: NCT06783777
Title: Study on the Correlation Between Tracheotomy Tip Pressure and Esophageal Pressure in Patients Weaned from Tracheotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: B2024-526R
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Distress Syndrome (RDS); Respiratory Ilness
Keywords: esophageal-pressure; tracheotomy tip pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Esophageal pressure monitoring — Esophageal pressure and Tracheotomy tip pressure were measured simultaneously in patients with off-line tracheotomy to verify the correlation
Device: Tracheotomy tip pressure — Esophageal pressure and tracheotomy tip pressure were measured simultaneously in patients with off-line tracheotomy to verify the correlation

SUMMARY:
Whether the correlation between gas incision tip pressure fluctuations (ΔPtt) and esophageal pressure fluctuations (ΔPes) is a potential measure of spontaneous respiratory effort in patients undergoing gas incision offline.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old), regardless of gender
* Tracheostomized patients with spontaneous breathing;
* Weaning criteria: under the condition of mask oxygen inhalation at 5L/min, SPO2 > 94%, PaO2/FiO2 > 150 - 200.
* The patient has stable hemodynamics and pH ≥ 7.32;
* Agree to participate in this trial and sign the informed consent form.

Exclusion Criteria:

* Patients with contraindications for esophageal catheter insertion and unable to monitor esophageal pressure;
* Patients with bleeding risks: severe coagulation disorders, esophageal varices；
* Local injuries: basilar skull fracture, maxillofacial fracture;
* Pregnant women;
* Patients considered not suitable by the researcher.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Correlation between esophageal pressure and tracheotomy tip pressure | 2 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital afraid of Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes